CLINICAL TRIAL: NCT03492437
Title: Phase I, Open-label, Single Sequence, Two-Period Study to Evaluate the Effect of Tepotinib on P-gp by Investigating the PK of the P-gp Probe Substrate Dabigatran Etexilate in Healthy Subjects
Brief Title: Effect of Tepotinib on the PK of the P-gp Substrate Dabigatran Etexilate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200095_0032; 2017-004074-34 (EudraCT Number)
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Results first posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: Non-small cell lung cancer (NSCLC); P-glycoprotein; Tepotinib; Dabigatran Etexilate
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Dabigatran; tepotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dabigatran Etexilate (Experimental)
  Interventions: Drug: Dabigatran Etexilate
- Tepotinib + Dabigatran (Experimental)
  Interventions: Drug: Dabigatran Etexilate; Drug: Tepotinib

INTERVENTIONS:
Drug: Dabigatran Etexilate — Participants received single oral dose of Dabigatran etexilate on Day 1 of Treatment period 1 and co-administration of Dabigatran with Tepotinib on Day 8 of Treatment period 2.
Drug: Tepotinib — Participants received single oral dose of Tepotinib for 8 days in Treatment period 2.
  Arms: Tepotinib + Dabigatran

SUMMARY:
This study investigated the effect of Tepotinib on the pharmacokinetics (PK) of the p-glycoprotein (P-gp) probe substrate Dabigatran etexilate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants of non-child bearing potential
* Body weight between 50 to 100 kilogram (kg)
* Body mass index (BMI) between 18.5 and 29.9 kilogram per meter square (kg/m^2)
* A male participant must agree to use and to have his female partner of childbearing potential to use highly effective method of contraception
* Participant must have given written informed consent before any study-related activities
* All values for hematology, coagulation, and biochemistry tests of blood and urinalysis are within the normal range. Minor (solitary) non-clinically relevant deviation(s) are allowed as judged by the Investigator
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participation in a clinical study within 60 days prior to first drug administration
* Whole blood donation or loss of > 450 milliliter (mL) within 60 days prior to first drug administration
* Any surgical or medical condition, or any other significant disease that could interfere with the study objectives, conduct, or evaluation
* Supine systolic blood pressure (SBP) greater than (>) 140 millimeter of mercury (mmHg) or less than (<) 90 mmHg, diastolic blood pressure (DBP) > 90 or < 50 mmHg, and pulse rate > 90 or <50 beats per minute (bpm) at Screening and at admission on Day-1.
* 12-Lead electrocardiograms (ECG) showing a corrected QT interval per Fridericia's formula (QTcF) > 450 milliseconds (ms), PR > 215 ms, or QRS > 120 ms (at Screening)
* Creatinine clearance estimated glomerular filtration rate (eGFR) < 90 milliliter per minute (mL/min) (at Screening)
* Participants with gall bladder removal or other relevant surgery of gastrointestinal tract
* History of any malignancy
* History of epilepsy
* Ascertained or presumptive allergy/hypersensitivity to the active drug substance and/or excipients
* Participants who in the Investigator's judgment were perceived as having an increased risk of bleeding
* Positive screen for alcohol or drugs of abuse (at Screening and Day -1)
* Positive screen for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV), and human immunodeficiency virus 1 and 2 antibodies (HIV1/HIV2 antibodies) (at Screening)
* Excessive consumption of xanthine-containing food or beverages before study drug administration until collection of last pharmacokinetic (PK) sample in each period (at Screening and Day -1)
* Receipt of any prescription or nonprescription medication within 14 days or 5 half-lives, before study drug administration
* Smoker or former smoker who stopped smoking less than 6 months before the time of the Screening Visit
* Intake of grapefruit, Seville orange, cranberry or juices of these 3 fruits, or St. John's Wort, from 14 days prior to Day -1
* Inability to communicate or cooperate with the Investigator
* Other factors, which in the opinion of the Investigator may interfere with study conduct (at Screening and Day -1 of first Period only)
* Legal incapacity or limited legal capacity
* Participants kept in detention
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

REFERENCES:
- [Derived] Yalkinoglu O, Becker A, Krebs-Brown A, Vetter C, Lupfert C, Perrin D, Heuer J, Biedert H, Hirt S, Bytyqi A, Bachmann A, Strotmann R. Assessment of the potential of the MET inhibitor tepotinib to affect the pharmacokinetics of CYP3A4 and P-gp substrates. Invest New Drugs. 2023 Aug;41(4):596-605. doi: 10.1007/s10637-023-01378-z. Epub 2023 Jul 6. PMID 37415001
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200095_0032
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html
- See also: Redacted Clinical study report, redacted clinical study protocol and redacted statistical analysis plan for this study is also available at the HC-PRCI portal (Health Canada-Public release of clinical information) — https://clinical-information.canada.ca/ci-rc/item/242300

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 39 participants were screened in this study. Out of which, 20 participants received Dabigatran and Tepotinib + Dabigatran treatment.
Groups:
- Dabigatran Etexilate: Participants received a single oral dose of 75 milligrams (mg) dabigatran etexilate capsule on Day 1 under fed state in treatment period 1.
- Tepotinib + Dabigatran: All participants who received 75 mg Dabigatran Etexilate in treatment period 1, received oral dose of 500 mg tepotinib film-coated tablets from Day 1 to 8 under fed state along with 75 mg dabigatran etexilate on Day 8 of treatment period 2.
Period: Treatment Period 1
Arm/Group | Dabigatran Etexilate | Tepotinib + Dabigatran
Started | 20 | 0
Completed | 20 | 0
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Dabigatran Etexilate | Tepotinib + Dabigatran
Started | 0 | 20
Completed | 0 | 19
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who received a single oral dose of 75 mg dabigatran etexilate capsule in treatment period 1 and 500 mg tepotinib (500 mg) film coated tablet from Day 1 to 8 along with 75 mg dabigatran etexilate Capsule in treatment period 2 under fed state.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under Plasma Concentration-time Curve From Time Zero to Last Sampling Time (Tlast) at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of Total Dabigatran
Description: AUC0-t was calculated according to the mixed log linear trapezoidal rule.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours Post-dose on Day 1 and Day 8
Population: Pharmacokinetic (PK) analysis set: all participants who completed at least 1 period without any relevant protocol violations with respect to factors affecting comparability of PK results with adequate study drug compliance and evaluable dabigatran PK data. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Dabigatran Etexilate | Tepotinib + Dabigatran
Number analyzed (Participants) | 20 | 19
nanogram*hour per milliliter (ng*h/mL) | 461 (74.9) | 709 (64.6)
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Tepotinib + Dabigatran; Test type: Other; Ratio of Geometric Least square Mean = 151.38, 90% CI 2-sided [127.35 to 179.93]

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Total Dabigatran
Description: AUC0-inf was calculated as AUC0-t plus (+) AUCextra. AUCextra represents the extrapolated part of AUC0-inf calculated by Clastpred/Lambda z, where Clastpred is the predicted plasma concentration at the last sampling time point, calculated from the log-linear regression line for Lambda z determination at which the measured plasma concentration is at or above Lower limit of quantification (LLOQ).
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours Post-dose on Day 1 and Day 8
Population: PK analysis set: all participants who completed at least 1 period without any relevant protocol violations with respect to factors affecting comparability of PK results with adequate study drug compliance and evaluable dabigatran PK data. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Dabigatran Etexilate | Tepotinib + Dabigatran
Number analyzed (Participants) | 19 | 19
ng*hr/mL | 544 (32.8) | 730 (61.8)
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Tepotinib + Dabigatran; Test type: Other; Ratio of Geometric Least square Mean = 144.70, 90% CI 2-sided [122.89 to 170.39]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Total Dabigatran
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours Post-dose on Day 1 and Day 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Dabigatran Etexilate | Tepotinib + Dabigatran
Number analyzed (Participants) | 20 | 19
Nanogram per milliliter (ng/mL) | 54.5 (72.8) | 76.9 (61.8)
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Tepotinib + Dabigatran; Test type: Other; Ratio of Geometric Least square Mean = 138.45, 90% CI 2-sided [121.59 to 157.65]

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Total Dabigatran
Description: Tmax is time to reach maximum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours Post-dose on Day 1 and Day 8
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour
Arm/Group | Dabigatran Etexilate | Tepotinib + Dabigatran
Number analyzed (Participants) | 20 | 19
Hour | 3.00 [1.50 to 6.00] | 4.00 [2.00 to 6.00]
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Tepotinib + Dabigatran; Test type: Other; Median Difference (Net) = 0.5, 90% CI 2-sided [-0.3 to 1.0]

5. Secondary Outcome: Elimination Half Life (t1/2) of Total Dabigatran
Description: Elimination Half Life (t1/2) was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours Post-dose on Day 1 and Day 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Dabigatran Etexilate | Tepotinib + Dabigatran
Number analyzed (Participants) | 19 | 19
Hour | 8.18 (12.9) | 7.81 (13.5)

6. Secondary Outcome: Apparent Clearance (CL/f) of Total Dabigatran
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours Post-dose on Day 1 and Day 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Dabigatran Etexilate | Tepotinib + Dabigatran
Number analyzed (Participants) | 19 | 19
Liter per hour (L/h) | 138 (32.8) | 103 (61.8)

7. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/f) of Total Dabigatran
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/f after oral dose was influenced by the fraction absorbed.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours Post-dose on Day 1 and Day 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Dabigatran Etexilate | Tepotinib + Dabigatran
Number analyzed (Participants) | 19 | 19
Liter | 1627 (34.7) | 1157 (58.4)

8. Secondary Outcome: Percentage of Area Under the Plasma Concentration-Time Curve From Time Tlast Extrapolated to Infinity (AUC0-inf) Obtained by Extrapolation (AUCextra%) of Total Dabigatran
Description: The AUC from time tlast extrapolated to infinity given as percentage of AUC0-inf. AUCextra% = (AUCextra /AUC0-inf)*100.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours Post-dose on Day 1 and Day 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC0-inf
Arm/Group | Dabigatran Etexilate | Tepotinib + Dabigatran
Number analyzed (Participants) | 20 | 19
percentage of AUC0-inf | 3.03216 (55.1249) | 2.3654 (63.8621)

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: Adverse event (AE) was defined as any untoward medical occurrence in participants which does not necessarily have causal relationship with treatment. AE was any unfavorable and unintended sign (including abnormal laboratory finding), symptom/disease temporally associated with use of medicinal product, whether/not considered related to medicinal product. A serious adverse event (SAE) was AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE is defined as AEs starting/worsening after first intake of the study drug. TEAEs included both serious TEAEs and non-serious TEAEs.
Time Frame: Screening up to Day 4 in Period 1; Day 1 up to Day 15 in Period 2
Population: The safety analysis set included all participants who received at least 1 dose of the planned investigational medicinal product (IMP).
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate | Tepotinib + Dabigatran
Number analyzed (Participants) | 20 | 20
Participants
  Treatment-emergent Adverse Events (TEAEs) | 4 | 15
  Serious TEAEs | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Values
Description: Number of participants with clinically significant change in laboratory values were reported. Clinical significance was decided by the investigator. Laboratory investigation included hematology, biochemistry, virology, drugs of abuse, hormones, urinalysis, and coagulation.
Time Frame: Screening up to Day 4 in Period 1; Day 1 up to Day 15 in Period 2
Population: The safety analysis set included all participants who received at least 1 dose of the planned IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate | Tepotinib + Dabigatran
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Changes in 12-lead Electrocardiogram (ECG) Findings
Description: Number of participants with clinically significant change in 12-lead ECG were reported. Clinical significance was decided by the investigator. The 12-lead ECGs were recorded after the participant have rested for at least 5 minutes in supine position.
Time Frame: Screening up to Day 4 in Period 1; Day 1 up to Day 15 in Period 2
Population: The safety analysis set included all participants who received at least 1 dose of the planned IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate | Tepotinib + Dabigatran
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Number of participants with clinically significant change in vital signs were reported. Clinical significance was decided by the investigator. Vital signs included body temperature, blood pressure, and pulse rate.
Time Frame: Screening up to Day 4 in Period 1; Day 1 up to Day 15 in Period 2
Population: The safety analysis set included all participants who received at least 1 dose of the planned IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate | Tepotinib + Dabigatran
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening up to Day 4 in Period 1; Day 1 up to Day 15 in Period 2
Arm/Group | Dabigatran Etexilate | Tepotinib + Dabigatran
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/20 | 15/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate (N=20) | Tepotinib + Dabigatran (N=20)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 7
Diarrhoea (Gastrointestinal disorders) | 1 | 11
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Faeces hard (Gastrointestinal disorders) | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 6
Tongue ulceration (Gastrointestinal disorders) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2
Heart rate increased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT03492437/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT03492437/SAP_001.pdf